CLINICAL TRIAL: NCT01448564
Title: Effects of Light-emitting Diodes (LED) on Peripheral Muscle Function, Exercise Tolerance and Cardiorespiratory Response During Exercise in Patients With Chronic Obstructive Pulmonary Disease
Brief Title: Effects of Laser Therapy on Muscle Function in COPD Patients
Acronym: LTCOPD
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Eduardo Foschini Miranda (Other)
Responsible Party: Sponsor-Investigator, Eduardo Foschini Miranda, Principal Investigator, University of Nove de Julho
Organization: University of Nove de Julho (Other)
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: COPD; COPD - LED (Other: COPD - LED)
Record Dates: First submitted 2011-10-03; First posted 2011-10-07 (Estimated); Last update posted 2013-09-04 (Estimated); Status verified 2013-09

CONDITIONS: Chronic Obstructive Pulmonary Disease; Fatigue
Keywords: Chronic Obstructive Pulmonary Disease; Fatigue; laser therapy
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive; Fatigue | interventions — Laser Therapy

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Laser therapy (Active Comparator): Recently has been using the LED, known by its acronym in English LED (Light Emitting Diode), devices that are light-emitting non-coherent and monochromatic, having a longer wavelength (± 10 - 30 nm) compared to lasers. The difference between the fundamental radiation emitted by a laser and an LED is the coherence of the beam.
  Interventions: Other: Laser therapy
- Placebo Laser therapy (Placebo Comparator)
  Interventions: Other: Placebo laser therapy

INTERVENTIONS:
Other: Laser therapy — The therapeutic effects of low intensity lasers are: (i) analgesic and anti-inflammatory, (ii) regeneration, (iii) tissue healing and (vi) recovery from muscle fatigue.
  Other Names: (Light Emitting Diode)
  Arms: Laser therapy
Other: Placebo laser therapy — The application of laser therapy will be a low intensity laser.
  Arms: Placebo Laser therapy

SUMMARY:
Light-emitting diodes (LEDs) have been used to minimize muscle fatigue in athletes and healthy subjects. Patients with chronic obstructive pulmonary disease (COPD) are susceptible to early muscle fatigue. The objective of this study is to assess the acute effects of LEDs on muscle function, exercise capacity, and cardiorespiratory responses during isometric and dynamic exercise in patients with COPD. This study will assess 30 patients with moderate to severe obstruction (FEV1 ≤ 70% predicted). Isometric and dynamic protocols will be conducted in two visits each, for a total of four visits a week a part. First, a venous blood sample will be taken from the patients. The isometric protocol will start with the determination of the maximum voluntary isometric contraction (MIVC) to determine the workload (60% of MIVC) for the isometric endurance test (IET). Patients will be randomized to receive either the placebo or LED application. Immediately after finishing this procedure, the patients will carry out the IET until the limit of tolerance or until a 20% fall of strength is observed. After the test, another blood sample will be taken. In the other visit (one week later), the same order of procedures will be performed, except with the opposite (LED or placebo). For the dynamic protocol, the same procedures described above will be followed except with the maximal incremental cycle ergometer test used instead of the IET. The electromyography will be recorded during the isometric and dynamic protocols. Differences in muscle function, exercise capacity, and cardiorespiratory responses between the LED and placebo applications will be analyzed. The therapeutic effects of LED could minimize muscle fatigue in patients with COPD by increasing exercise tolerance.

ELIGIBILITY:
Inclusion Criteria:

* 35 patients will be selected (see sample calculation in Section 6) who have moderate to severe obstruction (FEV1 ≤ 70% predicted) and stable disease, as suggested by the absence of changes in medication in the last 4 weeks.

Exclusion Criteria:

* Ischemic heart disease, recent surgery, neuro-muscular or orthopedic that limit the performance of the protocol.
* Patients will only be included in the study after signing the consent form.

Ages: 40 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 27 (Estimated)
Dates: Start 2012-06; Primary Completion 2013-12; Study Completion 2013-12

PRIMARY OUTCOMES:
Analysis of the recovery time for the isometric and dynamic protocol | Measures muscular endurance will be compared after a period of 1 week.

SECONDARY OUTCOMES:
Analysis of lactate levels and the activity of CK and C-reactive protein (CRP). | Measures blood will be compared after a period of 1 week.

CONTACTS AND LOCATIONS:
Overall Officials: Eduardo Miranda, Principal Investigator
Locations (1):
- University Nove de Julho, São Paulo, São Paulo, Brazil

REFERENCES:
- [Derived] Miranda EF, Leal-Junior EC, Marchetti PH, Dal Corso S. Effects of light-emitting diodes on muscle fatigue and exercise tolerance in patients with COPD: study protocol for a randomized controlled trial. Trials. 2013 May 10;14:134. doi: 10.1186/1745-6215-14-134. PMID 23663518